CLINICAL TRIAL: NCT06963229
Title: Cognitive Changes After Hip Prosthesis; Comparison Between Combined Lumbosacral Nerve Block Versus Spinal Anesthesia: A Double Blind Randomized Clinical Trial
Brief Title: Spinal Anesthesia Vs. Neve Block in Risk of Cognitive Decline
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Omar Rajab, Chairman of Anesthesia Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MGH-07-24002
Record Dates: First submitted 2025-04-21; First posted 2025-05-08 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Cognitive Complications
Keywords: Fractures, Hip; Nerve Block; Spinal Anesthesia; Nerve, Sciatic; paravertebral; Aged
MeSH Terms: conditions — Postoperative Cognitive Complications; Hip Fractures | interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Anesthesia (Active Comparator)
  Interventions: Procedure: Spinal Anesthesia (bupivacaine)
- Lumbosacral Nerve Block (Active Comparator)
  Interventions: Procedure: Peripheral Nerve Block

INTERVENTIONS:
Procedure: Spinal Anesthesia (bupivacaine) — L3-L4 or L4-L5 3cc of 2% bupivacaine
  Arms: Spinal Anesthesia
Procedure: Peripheral Nerve Block — Sciatic Nerve Block 20ml of Anesthetic Mixture, Paravertebral Nerve Block (L3-L4 and L4-L5) 20ml of Anesthetic Mixture
  Mixture Details:
  * 5ml Lidocaine 2%
  * 5ml Lidocaine 1% with Adrenaline (1-200000)
  * 10ml Bupivacaine 0.5%
  Arms: Lumbosacral Nerve Block

SUMMARY:
Hip fracture is a potentially devastating event, and serious surgical and medical complications occur frequently especially for elderly patients. Delirium is one of the common complications after hip surgery.

This study objective is to assess the association between type of anesthesia (nerve block vs. spinal anesthesia) and risk of cognitive decline (CD). And its secondary objective is to compare intra-operative hemodynamic changes, and post-operative pain.

Prospective, double blind randomized clinical trial of hip fracture patients who will be assessed for CD pre- and postoperatively, for three months after surgery. Patients undergoing hip surgery will be randomized into two groups. Group 1 will receive unilateral lumbosacral nerve block (sciatic nerve block and paravertebral block at levels L3-L4 and L4-L5) as well as placebo injection (1 ml normal saline) at the spinal anesthesia level (L3-L4 or L4-L5). Group 2 will receive spinal anesthesia in addition to placebo injection at the sciatic, L3-L4 and L4-L5 levels.

DETAILED DESCRIPTION:
Hip fracture is a potentially devastating event, and serious surgical and medical complications occur frequently especially for elderly patients. Around one-third of the patients pass away within the first post-operative year.

One of the most common complications in hip fracture patients is delirium which is characterized by an acute disturbance in awareness, attention and cognitive function. Delirium has a fluctuating course and is usually reversible. However, evidence suggests an association between delirium and future cognitive decline and development of dementia during months after the delirium episode. Dementia is a chronic syndrome characterized by cognitive decline, impairment in activities of daily living and a change in social abilities and behavior.

Several risk factors are identified for preoperative and postoperative delirium including age, comorbidities, intraoperative hypotension and use of vasopressors. There is some controversy about the cognitive consequences due to the type of anesthesia used.

Spinal and general anesthesia are commonly used for hip surgery. An alternative technique is the combined sciatic-paravertebral block that has been used to overcome the adverse effects associated with spinal and general anesthesia. This anesthetic technique was associated with less intraoperative hypotension and reduced rate of ICU admission. Given the promising effect of paravertebral block on the outcome of hip surgery, we will conduct this study to assess the effect of paravertebral block on postoperative CD.

ELIGIBILITY:
Inclusion Criteria:

* Admitted with a hip fracture (femoral neck, trochanteric or sub-trochanteric)
* 65 years or older
* 40 Kgs in weight and higher

Exclusion Criteria:

* Uncooperative
* Considered as moribund by the orthopedic surgeon at admission
* Alzheimer
* Severe cognitive impairment (MMSE<18)
* Absolute contraindication for spinal anesthesia (assessed preoperatively)
* Allergy to local anesthesia
* Have any severe visual disorder or debilitating vascular event

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Cognitive Decline Post-operatively | 3 Months
  A questionnaire will be used to collect data. Demographic information including age (by year), gender, ASA score (I-IV), BMI (kg/m^2), clinical condition pre-fracture (MMSE Score), as well as type and duration (by days) of fracture will be collected. The patient's cognitive function will be assessed before the operation using the MMSE. The MMSE is a validated questionnaire that is comprised of six sections examining the following functions: orientation, registration, attention and calculation, recall, language, as well as ability to follow simple commands and orientation.
  Illiterate patients will not be asked the questions pertaining to attention and calculation in addition to language questions. Hence, for these patients the score will be over 23 but it will be converted to a score over 30.
  Total Score is 30; a score between 24 and 30 indicates no cognitive impairment, a score between 18 and 23 means mild cognitive impairment and a score between 0 and17 indicates severe impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naja Z, el Hassan MJ, Khatib H, Ziade MF, Lonnqvist PA. Combined sciatic-paravertebral nerve block vs. general anaesthesia for fractured hip of the elderly. Middle East J Anaesthesiol. 2000 Jun;15(5):559-68. PMID 11126507
- [Background] Zywiel MG, Prabhu A, Perruccio AV, Gandhi R. The influence of anesthesia and pain management on cognitive dysfunction after joint arthroplasty: a systematic review. Clin Orthop Relat Res. 2014 May;472(5):1453-66. doi: 10.1007/s11999-013-3363-2. PMID 24186470
- [Background] Davis N, Lee M, Lin AY, Lynch L, Monteleone M, Falzon L, Ispahany N, Lei S. Postoperative cognitive function following general versus regional anesthesia: a systematic review. J Neurosurg Anesthesiol. 2014 Oct;26(4):369-76. doi: 10.1097/ANA.0000000000000120. PMID 25144505
- [Background] Tzimas P, Samara E, Petrou A, Korompilias A, Chalkias A, Papadopoulos G. The influence of anesthetic techniques on postoperative cognitive function in elderly patients undergoing hip fracture surgery: General vs spinal anesthesia. Injury. 2018 Dec;49(12):2221-2226. doi: 10.1016/j.injury.2018.09.023. Epub 2018 Sep 11. PMID 30526923
- [Background] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Abrahamsen B, van Staa T, Ariely R, Olson M, Cooper C. Excess mortality following hip fracture: a systematic epidemiological review. Osteoporos Int. 2009 Oct;20(10):1633-50. doi: 10.1007/s00198-009-0920-3. Epub 2009 May 7. PMID 19421703
- See also: Related Info — https://doi.org/10.1186/1741-7015-12-63
- See also: Related Info — https://books.google.com.lb/books?hl=en&lr=&id=Tw5eAtsatiUC&oi=fnd&pg=PA1&dq=World+Health+Organization.+ICD-10:+International+classification+of+diseases+and+related+health+problems,10th+Rev.ed.+New+York,+NY:+World+Health+Organization%3B+2008.&ots=o5b0hYpGqK&sig=avE0Te1tTONYq1kyWBzeo1TCKTE&redir_esc=y#v=onepage&q&f=false